CLINICAL TRIAL: NCT02041039
Title: Reward System Responses to Food Aromas
Status: Completed | Type: Observational
Sponsor: Robert Considine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Robert Considine, Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: R01DK089070 (NIH)
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum/plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal weight: non-smoking, right handed women age 18-40 years BMI between 18-25 kg/m2
- overweight/obese: non-smoking, right-handed women age 18-40 year BMI 30-50 kg/m2 (maximum weight 350 pounds, shoulder width no greater than 23/5 inches)

SUMMARY:
Food aromas are a part of foods' flavor, and can promote overeating. Alcohol consumption also stimulates appetite, and contributes to overeating while under alcohol's acute effects. Knowing the brain regions that respond to food aromas and alcohol, and how they are modified by the amount of body fat and alcohol exposure, will provide critical information about the neural systems that underlie loss of control of eating. Therefore, the main hypotheses of this study are that: A) Lean and obese subjects have different brain responses to food aromas that enhance desire to eat, and B) Acute alcohol intoxication i) enhances the brain's response to food odors, and ii) affects brain systems that inhibit or terminate eating. To test these hypotheses, we have modified functional magnetic resonance imaging (fMRI) paradigms successfully used to study alcoholic drink aromas in subjects at risk for alcoholism.

DETAILED DESCRIPTION:
Food aromas are powerful appetitive cues that are intrinsic to foods' flavor and hedonic qualities, and such cues can facilitate overeating. Alcohol consumption similarly "primes" appetite, and contributes to overeating while under alcohol's acute effects. Knowing the brain loci that respond to such naturalistic appetitive stimuli, and how they are modified by body fat and alcohol exposure, will provide critical insights about the neural systems that underlie loss of control of eating. Therefore, the main hypotheses of this study are that: A) Lean and obese subjects have different limbic responses to the olfactory cues that enhance motivation to eat, and B) Acute alcohol intoxication i) potentiates the brain's reward system response to food odors, and ii) affects brain systems involved in behavioral inhibition and eating restraint. To test these hypotheses, we have modified functional magnetic resonance imaging (fMRI) paradigms successfully used to study alcoholic drink aromas in subjects at risk for alcoholism.

ELIGIBILITY:
Inclusion Criteria:

* non smoking, right handed women 18-40 years
* good health without self reported neurological or psychiatric disorder
* no indication of eating disorders
* normal sense of smell

Exclusion Criteria:

* pregnant,/breast feeding women
* history of drug abuse/dependence, positive drug screen for amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates or PCP
* DSM-IV axis I psychiatric disorders or head injury with loss of consciousness
* contraindications to MRI (ferrous material, claustrophobia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: subjects to be drawn from the Indianapolis and greater metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2011-04-15 (Actual); Primary Completion 2015-09-11 (Actual); Study Completion 2015-09-11 (Actual)

PRIMARY OUTCOMES:
neural response to food odor | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Eiler WJ 2nd, Dzemidzic M, Case KR, Armstrong CL, Mattes RD, Cyders MA, Considine RV, Kareken DA. Ventral frontal satiation-mediated responses to food aromas in obese and normal-weight women. Am J Clin Nutr. 2014 Jun;99(6):1309-18. doi: 10.3945/ajcn.113.080788. Epub 2014 Apr 2. PMID 24695888